CLINICAL TRIAL: NCT05298618
Title: Magnesium Administration After Cardioplegic Arrest With Del Nido Cardioplegia
Acronym: MGSO
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0816
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Del Nido Cardioplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All patients undergoing CPB with dNC cardioplegic arrest shall have two magnesium levels measured. The first sample shall be taken prior to magnesium administration and within 30 minutes of cross-clamp removal. The second sample will be drawn 10 +/- 5 minutes after cross-clamp removal and magnesium administration. Magnesium levels will be analyzed and compared against normally expected values.

SUMMARY:
The cardioplegia solution of choice in many pediatric cardiac congenital programs is the del Nido solution. While many cardioplegia solutions provide diastolic arrest, del Nido provides a longer period of time between doses of cardioplegia. Many of the other cardioplegia solutions do not incorporate magnesium into the constituents, but del Nido does. Routine practice at CCHMC is to dose 25 mg/kg magnesium upon removal of the heart cross-clamp to protect against hypomagnesemia and associated arrhythmias. However, with the incorporation of magnesium in the del Nido solution, it may not be necessary to administer magnesium post cross-clamp and it could in fact be detrimental if the magnesium level is too high. This observational study will examine the magnesium levels prior to and after cross-clamp removal under our current process. The magnesium levels measured after the administration of del Nido cardioplegia and prior to cross-clamp removal will help inform our current practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery requiring CPB and cardioplegic arrest with del Nido cardioplegia solution.
* Patients planned to receive post cross-clamp dose of 25 mg/kg magnesium sulfate.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing CPB with dNC cardioplegic arrest.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Examine magnesium levels prior to and after cross-clamp. | 24 months from start of enrollment.
  The primary objective of this study is to examine magnesium levels prior to and after cross-clamp.

CONTACTS AND LOCATIONS:
Overall Officials: James Reagor, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided